CLINICAL TRIAL: NCT05160272
Title: Effects of GABAA Receptor Modulation by AP-325 on Insulin
Brief Title: Effects of GABAA Receptor Modulation by AP-325 on Insulin Secretion in Patients with Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Deutsche Diabetes Forschungsgesellschaft e.V. (Other)
Collaborators: Algiax Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Organization: German Diabetes Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GAP-325
Record Dates: First submitted 2021-11-17; First posted 2021-12-16 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Type2 Diabetes
Keywords: Type 2 Diabetes; Diabetes mellitus; GABAA receptor; β-cell function; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AP-325 Treatment (Experimental): AP-325, film-coated tablet, 50mg once daily
  Interventions: Drug: AP-325
- Placebo Treatment (Placebo Comparator): Placebo matching AP-325 film-coated tablet, once daily
  Interventions: Drug: Placebo matching AP-325

INTERVENTIONS:
Drug: AP-325 — Measurement of the effect of AP-325 50mg/d compared to matching placebo after 4-week treatment.
  Arms: AP-325 Treatment
Drug: Placebo matching AP-325 — Measurement of the effect of AP-325 50mg/d compared to matching placebo after 4-week treatment.
  Arms: Placebo Treatment

SUMMARY:
The aim of this single-center, prospective, randomized, double-blind, placebo-controlled, 2-arm parallel-group interventional study is to investigate the effect of 4-week treatment with AP-325 on C-peptide release as measure of insulin secretion compared to placebo in type 2 diabetes (T2D) patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2D
* Age between 25 and 75 years
* HbA1c ≥6.5 and ≤9.5 %
* BMI ≤ 45 kg/m2
* Treatment-naive or stable antihyperglycemic therapy with metformin, α-glucosidase-inhibitor and/or SGLT2 inhibitor
* Ability to give consent

Exclusion Criteria:

* Acute infections (hsCRP > 5mg/dl, body temperature >37.5°C)
* Insulin therapy or treatment with sulfonylureas, glinides, GLP-1 receptor agonists, thiazolidinediones; current treatment with DPP-4 inhibitors or during the 4 weeks prior to baseline examination
* Uncontrolled hyperglycemia, e.g. fasting blood glucose >240 mg/dl
* Heart rate <50 or >100 beats per minute; systolic blood pressure <100 or >160 mmHg; diastolic blood pressure <50 or >100 mmHg; uncontrolled hypertension
* Creatinine clearance <60 ml/min (eGFR by MDRD formula)
* Severe chronic illnesses, such as congestive heart failure (NYHA III/IV), liver insufficiency (Child-Pugh Class B/C), history of acute coronary syndrome, stroke
* Anemia (Hb <12 g/l for men, Hb <11 g/l for women)
* Participation in another intervention study within 2 months before the examination
* Hypersensitivity against AP-325, placebo or other ingredients of IMP
* Immunocompromising diseases
* Immunomodulatory drugs (e.g. oral cortisone preparations, biologicals)
* Thyroid diseases with an unstable metabolic state (change in L-thyroxine dose within the past 6 weeks, TSH and fT4 outside the normal range)
* Planned pregnancy, pregnant or lactating women, positive pregnancy test, and woman of childbearing potential not using two adequate methods of contraception, including a barrier method and a highly efficacious non-barrier method
* Past (≤ 5 years) or current history of psychiatric disorders, including psychiatric depression
* HIV, hepatitis B or C disease
* Previous / current alcohol and / or drug abuse
* Malignant cancer
* BIA and MR-incompatible metal or magnetic implants, devices or objects inside of or on the body, claustrophobia
* Treatment with the following drug groups or agents:

Anticoagulant drugs (exception: acetylsalicylic acid 100 mg/day), dihydropyridines (e.g. nifedipine, amlodipine), azilsartan, losartan and irbesartan, celecoxib; if applicable, other drugs that are predominantly metabolized by CYP2C9

* Inhibitors or inducers of CYP2C9, CYP3A4, such as amiodarone, verapamil, rifampicin
* Poor CYP2C9 metabolizer

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Circulating C-peptide by iAUC of C-peptide during an IVGTT | 4 weeks
  Change in circulating C-peptide levels from baseline to end of intervention measured by iAUC of C-peptide during an IVGTT until 60th minute (second phase) with AP-325 compared to placebo

SECONDARY OUTCOMES:
Basal insulin level | 4 weeks
  Change in basal insulin level from baseline to end of treatment
C-peptide level | 4 weeks
  Change in C-peptide level from baseline to end of treatment
Glucose level | 4 weeks
  Change in glucose level from baseline to end of treatment
iAUC of circulating insulin (overall) | 4 weeks
  Change in iAUC of circulating insulin during an IVGTT from baseline to end of treatment
iAUC of C-peptide level (overall) | 4 weeks
  Change in C-peptide level during an IVGTT from baseline to end of treatment
iAUC of glucose level (overall) | 4 weeks
  Change in iAUC of glucose level during an IVGTT from baseline to end of treatment
iAUC of circulating insulin (AIR) (first 10 min) | 4 weeks
  Change in iAUC of circulating insulin (AIR) during an IVGTT in the first 10 minutes from baseline to end of treatment
iAUC of C-peptide (first 10 min) | 4 weeks
  Change in iAUC of C-peptide during an IVGTT in the first 10 minutes from baseline to end of treatment
iAUC of glucose (first 10 min) | 4 weeks
  Change in iAUC of glucose during an IVGTT in the first 10 minutes from baseline to end of treatment
disposition index (DI) | 4 weeks
  Change in the disposition index (DI) through Minimal Model during an IVGTT from baseline to end of treatment
peak insulin response | 4 weeks
  Change in peak insulin response during an IVGTT from baseline to end of treatment
insulin secretion rate (ISR) | 4 weeks
  Change in insulin secretion rate (ISR) during an IVGTT from baseline to end of treatment
fructosamine levels | 4 weeks
  Change in 1.5-Anhydroglucitol glucose from baseline to end of treatment
fructosamine levels II | 4 weeks
  Change in fructosamine level from baseline to end of treatment
fructosamine levels III | 4 weeks
  Change in fasting blood glucose from baseline to end of treatment
Plasma concentrations of AP-325 | 4 weeks
  Change in Plasma concentrations of AP-325 at 1 hour post-dose on Days 1 and 28; pre-dose on Days 4 and 28. Accumulation of Ctrough from Day 4 to Day 28
Ctrough-ss (Day 28) and the change from baseline to Day 28 | 4 weeks
  Change in relationship between Ctrough-ss (Day 28) and the change from baseline to Day 28 in primary and secondary endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, MD, Principal Investigator — Deutsches Diabetes-Zentrum
Locations (1):
- German Diabetes Center, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No